CLINICAL TRIAL: NCT00265889
Title: Tandem Autologous Stem Cell Transplantation for Patients With Primary Progressive or Poor Risk Recurrent Hodgkin's Disease
Brief Title: Autologous Stem Cell Transplant in Treating Patients With Progressive or Recurrent Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCF5386; P30CA043703 (NIH); CCF-5386 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Results first posted 2013-08-26 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-10

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Filgrastim; Busulfan; Cyclophosphamide; Etoposide; Melphalan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Poor Risk (Experimental): Primary progressive, recurrent, or resistant relapse patients
  Interventions: Biological: filgrastim; Drug: busulfan; Drug: cyclophosphamide; Drug: etoposide; Drug: melphalan; Procedure: autologous-autologous tandem hematopoietic stem cell transplantation; Radiation: radiation therapy
- Good Risk (Experimental): First recurrence patients
  Interventions: Biological: filgrastim; Drug: busulfan; Drug: cyclophosphamide; Drug: etoposide; Drug: melphalan; Procedure: autologous-autologous tandem hematopoietic stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — 480 mcg beginning day +5
Drug: busulfan — 11.2 mg/kg; 0.8 mg/kg IV q6h X 14 doses
Drug: cyclophosphamide — 60 mg/kg IV over 2 hours x 2 days
Drug: etoposide — 60 mg/kg, IV
Drug: melphalan — 150mg/m2 in NS at a concentration of 0.4mg/cc infused over 60 minutes.
Procedure: autologous-autologous tandem hematopoietic stem cell transplantation — autologous-autologous tandem hematopoietic stem cell transplantation
Radiation: radiation therapy — radiation therapy

SUMMARY:
RATIONALE: Giving two autologous stem cell transplants (one after the other) may be an effective treatment for Hodgkin's lymphoma.

PURPOSE: This phase II trial is studying how well giving two autologous stem cell transplants works in treating patients with progressive or recurrent Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 3-year progression-free survival of patients with progressive or recurrent Hodgkin's lymphoma treated with tandem autologous stem cell transplantation (2 courses of high-dose therapy with autologous stem cell rescue).
* Determine the response rate in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a pilot study. Patients are stratified according to risk (poor risk [primary progressive, recurrent, or resistant relapse] vs good risk [first recurrence]).

* Salvage therapy (for patients with relapsed disease after achieving a previous complete response): Patients receive at least 2 courses of salvage chemotherapy or radiotherapy.
* Autologous hematopoietic stem cell collection: Patients undergo autologous hematopoietic stem cell collection. Patients with an inadequate number of collected stem cells are removed from the study.
* First preparative regimen: Patients receive high-dose melphalan IV continuously over 16 hours on day -1.
* First autologous stem cell transplantation (SCT): Patients undergo autologous SCT on day 0. They also receive filgrastim (G-CSF) IV over 30 minutes once daily beginning on day 5 and continuing until blood counts recover. At least 4-8 weeks later, patients proceed to second preparative regimen.
* Second preparative regimen: Patients receive high-dose carmustine IV over 1-2 hours on days -6, -5, and -4, etoposide IV over 4 hours on day -3, and cyclophosphamide IV over 2 hours on day -2. Beginning 36-48 hours later, patients proceed to the second autologous SCT (day 0).
* Second autologous SCT: Patients undergo second autologous SCT on day 0. Patients also receive filgrastim (G-CSF) IV over 30 minutes once daily beginning on day 5 and continuing until blood counts recover.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* confirmed Hodgkin's lymphoma meeting ≥ 1 of the following criteria:

  * Disease progression during initial first line chemotherapy
  * Complete response lasting ≤ 90 days after induction
  * Partial response lasting ≤ 90 days after induction
  * First recurrence/progression with the duration of initial response ≤ 12 months after completion of chemotherapy NOTE: *There must be unequivocal radiological evidence of recurrent or progressive disease if biopsy was not obtained at time of disease recurrence/progression
* No clonal abnormalities in marrow collection
* Must have bilateral or unilateral bone marrow aspirates and biopsy within 42 days prior to stem cell collection
* Must have adequate sections of original diagnostic specimen available for review

  * Needle aspirations or cytologies are not adequate
* No prior lymphoma, myelodysplastic syndromes, or leukemia (even if disease free ≥ 5 years)
* No CNS involvement

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 50-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal* (ULN) NOTE: *Unless due to Hodgkin's lymphoma

Renal

* Creatinine clearance ≥ 60 mL/min
* Creatinine ≤ 2.0 times ULN

Cardiovascular

* Ejection fraction ≥ 45% by 2-D echocardiogram
* No significant active cardiac disease

Pulmonary

* Adequate pulmonary function
* DLCO ≥ 45%

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer
* No known HIV or AIDS infection
* No active bacterial, fungal, or viral infection
* No medical condition that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Chemotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2002-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Bolwell, MD, Study Chair — Cleveland Clinic Taussig Cancer Institute
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from medical clinic from August 2002 thru October 2010.
Pre-assignment Details: Only Poor Risk Patients were enrolled.
Groups:
- Poor Risk Patients: Poor Risk (primary progressive, recurrent, or resistant relapse)
Period: Overall Study
Arm/Group | Poor Risk Patients
Started | 42
Cycle 1: 1st Regimen/Transplant | 37
Cycle 2: 2nd Regimen/Transplant | 37
Completed | 37
Not Completed | 5
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Insurance denied the request | 3

BASELINE CHARACTERISTICS:
Arm/Group | Poor Risk Patients
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Outcome is based on the number of patients who were alive without progression or relapse within 1 year. Progression is defined as a 50% increase in the sum of products of all measurable lesions.
Time Frame: one year after second transplant
Population: Analysis is per protocol, so includes patients who received both transplants
Measure: Number; unit: participants
Arm/Group | Poor Risk Patients
Number analyzed (Participants) | 37
participants | 18

2. Primary Outcome: Response Rate
Description: Number of patients that receive a Complete Response (CR), Partial Response (PR)or Progression. CR defined as complete disappearance of all measurable and evaluable disease and no new lesions. PR is defined as >/= 50% decrease in the sum of products of all measurable lesions. Progression is defined as a 50% increase in the sum of products of all measurable lesions.
Time Frame: One year after second transplant
Population: Analysis is per protocol, so includes patients who received both transplants
Measure: Number; unit: participants
Arm/Group | Poor Risk Patients
Number analyzed (Participants) | 37
participants
  Complete Response | 18
  Progression | 14
  Unknown | 2
  Expired | 3
  Partial Response | 0

3. Primary Outcome: Number of Patients That Experience Pulmonary Toxicity
Description: Pulmonary toxicity are due to side effects that medicinal drugs cause to the lungs.
Time Frame: One year after second transplant
Population: Analysis is per protocol, so includes patients who received treatment
Measure: Number; unit: participants
Arm/Group | Poor Risk Patients
Number analyzed (Participants) | 37
participants | 9

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the patient went on study to off study, approximately a 6 month time frame per patient.
Arm/Group | Poor Risk Patients
Serious Adverse Events (participants affected / at risk) | 1/37
Other Adverse Events (participants affected / at risk) | 23/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Poor Risk Patients (N=37)
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Poor Risk Patients (N=37)
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 8
Cardiac Dysfuntion (Cardiac disorders) | 4
Fever (General disorders) | 5
Infections (Infections and infestations) | 11
Respiratory Dysfunction (Respiratory, thoracic and mediastinal disorders) | 3
Acute Renal Failure (Renal and urinary disorders) | 1
Gastrointestinal-other (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No